CLINICAL TRIAL: NCT01600547
Title: Odense Fallers and Osteoporosis Study
Acronym: OFOS
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Katja Thomsen, ph.d.student, University of Southern Denmark
Other Study IDs: s20110162
Record Dates: First submitted 2012-05-08; First posted 2012-05-17 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Accidental Falls; Osteoporosis; Disability
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- fall clinic population: women, aged + 65 years
- control fallers: randomly selected community aged matched female controls with a fall episode
- control non fallers: randomly selected community aged matched female controls, with out fall episodes

SUMMARY:
Osteoporosis and falls occur with increasing frequency among the elderly. Osteoporosis and fall increases the risk of fracture. Falls in the elderly are associated with a high morbidity and mortality with potentially life-threatening consequences of falls including fractures. Besides fracture fall may cause long term problems such as disability fear of falling and loss of independence. Today osteoporosis is diagnosed by bone scan of the hip and spine. The investigators want to investigate whether other more accessible and less expensive testing methods can be used to diagnose osteoporosis. Additionally, the investigators will examine the incidence of osteoporosis among the elderly in the municipality of Odense. Finally, the investigators would like to investigate the association between factors that can lead to falls and to investigate the performance of older and whether there are changes in functional ability over time.

DETAILED DESCRIPTION:
Study Objectives

1. To define the prevalence of osteoporosis in a falls clinic population, and compare it with two aged matched control groups - fallers not attending the falls clinic and non-fallers.
2. To evaluate the usefulness of peripheral bone scanning techniques in a falls clinic population.
3. To determine the prevalence of vertebral fractures in a falls clinic population and compare it with two aged matched control groups - fallers not attending the falls clinic and non-fallers
4. To investigate functioning, disability, health related quality of life and perceived need for rehabilitation in a falls clinic population including variation in a one year period, and compare it with two aged matched control groups - fallers not attending the falls clinic and non-fallers.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 65 years or over attending the falls clinic

  *(There will be no upper age limit to recruitment).
* Those capable of giving Informed consent.

Exclusion Criteria:

* Patients under the age of 65 years.
* Men.
* Patients unwilling to give informed consent.
* Cognitively impaired people who are not capable of giving consent.
* Patients who are not mobile enough to be helped onto a DXA scan table with help

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Consecutive patients attending the Odense University hospital falls clinic will be recruited to the study Two control groups will be recruited. A questionnaire will be sent to randomly selected community aged matched female controls.
Sampling Method: Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Bone mineral density using DXA of hip and spine regions (Hologic machine) | baseline
Prevalence of vertebral fractures using instant vertebral assessment mode (IVA) of the DXA machine (Hologic machine) | baseline
Bone mineral density of the phalanges using radiographic absorptiometry (Alara Metriscan machine) | baseline
Broad band ultrasound attenuation of the heel using the heel ultrasound machine (Lunar Achilles machine) | baseline
Fall incidences | one year
Mental health state | one year
  Meausered by Mini Mental State Examination (MMSE)
Health related quality of life | one year
  Self Reporting Questionnaire will be used
Perceived need | one year
  Self Reporting Questionnaire
Basis mobility | One year
  Time up and go, Chair stand, Bergs balance scale, Avlunds scale, gait speed and dual-task will be used
Fear of falling | One year
  The Falls Efficacy scale - international will be used
Muscle strength in upper and lower extremities | One year
  A dynamometer will be used

CONTACTS AND LOCATIONS:
Overall Officials: Katja Thomsen, MD, Principal Investigator — University of Southern Denmark; Lisbeth Rosenbek Minet, ph.d., Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital Geriatric department, Odense C, Denmark

REFERENCES:
- [Derived] Thomsen K, Ryg J, Matzen L, Hermann AP, Masud T. Choice of osteoporosis guideline has important implications for the treatment decision in elderly women referred to a fall clinic. Dan Med J. 2014 Dec;61(12):A4980. PMID 25441734